CLINICAL TRIAL: NCT07297706
Title: Pilates Exercises Versus Mirror Therapy on Shoulder Dysfunction Post Neck Dissection Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Yasmen gamal Elrakhawi, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Yasmen-Msc
Record Dates: First submitted 2025-12-09; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Pilates Exercise; Mirror Therapy; Shoulder Pain; Dissection
MeSH Terms: conditions — Shoulder Pain | interventions — Exercise Movement Techniques; Mirror Movement Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pilates exercises (Experimental): This group will include 26 patients suffering from shoulder post-neck dissection surgeries (Modified radical and selective NDS). They will receive the pilate exercises for 40 min/session, 3 sessions/ week for 8 weeks, in addition to the traditional physical therapy program (ROM exercises, pendulum exercises, shoulder wheel exercises, stretching, and strengthening exercises for shoulder muscles)
  Interventions: Other: Pilates exercises; Other: Traditional physical therapy
- Mirror therapy (Active Comparator): This group will include 26 patients suffering from shoulder dysfunction post neck dissection surgeries (modified radical, and selective NDS), they will receive Mirror therapy for 40 min/session, 3 sessions/ week for 8 weeks in addition to the traditional physical therapy program (ROM exercises, pendulum exercises, shoulder wheel exercises, stretching, and strengthening exercises for shoulder muscles)
  Interventions: Other: Mirror therapy; Other: Traditional physical therapy

INTERVENTIONS:
Other: Pilates exercises — Pilates exercise aids in recovery post-breast cancer surgery by improving daily living activities, shoulder function, and quality of life. It emphasizes principles such as centralization, concentration, control, precision, flow, and breathing, enhancing muscle strength and flexibility. Additionally, mild stretching exercises contribute to maintaining and increasing range of motion, and Pilates can be tailored to individual patient needs and abilities.
  Arms: Pilates exercises
Other: Mirror therapy — Mirror therapy has been shown to enhance shoulder function in patients with shoulder problems immediately after the intervention. Three-minute of Mirror therapy improved forward flexion by 14.5° in patients with shoulder pain and limited shoulder range of motion
  Arms: Mirror therapy
Other: Traditional physical therapy — including (ROM exercises, pendulum exercises, shoulder wheel exercises, stretching, and strengthening exercises for shoulder muscles)

SUMMARY:
The purpose of this study is to compare the therapeutic effects of pilates exercises and mirror therapy on shoulder dysfunction post-neck dissection surgeries.

DETAILED DESCRIPTION:
Shoulder morbidity is a significant concern for patients undergoing neck dissection in head and neck cancer treatment, with more extensive surgeries correlated with higher postoperative shoulder issues. Preservation of the spinal accessory nerve during modified radical neck dissection reduces shoulder dysfunction. Shoulder pain often results from trapezius deficits due to nerve injury, leading to symptoms like shoulder droop and loss of function. Current management of oral and oropharyngeal carcinoma focuses on selective procedures that maintain nonlymphatic structures in the neck, as extended dissections are linked to increased shoulder dysfunction. This study aims to compare the effectiveness of pilates exercises and mirror therapy in improving shoulder dysfunction after neck dissection surgeries.

ELIGIBILITY:
Inclusion Criteria:

1. Patient's age ranged between 35-55 years.
2. Both genders will participate in the study.
3. All patients suffering from shoulder dysfunction post-unilateral neck dissection surgeries ( modified radical and selective neck dissection surgeries).
4. All patients will have shoulder pain, limited ROM (flexion, abduction, external rotation) and limited shoulder function.
5. All patients will begin the treatment program 1-3 months after neck dissection surgeries.
6. All patients enrolled in the study will have their informed consent.

Exclusion Criteria:

1. Subjects suffering from active malignant tumors.
2. Subjects with rotator cuff tears or other shoulder ligaments injuries.
3. A history of neck or ipsilateral shoulder injuries, pain in the last 6-month prior neck dissection surgeries.
4. Adhesive capsulitis secondary to diabetes mellitus or fractures.
5. Recurrent shoulder dislocation.
6. Recent fractures or surgeries in the shoulder.
7. Neurological disorder
8. The presence of residual local regional cancer or distant metastases to other regions.
9. Comorbid medical illness or psychiatric illness and visual disturbance that would prevent completion of treatment.

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-09-13 (Actual); Study Completion 2025-10-13 (Actual)

PRIMARY OUTCOMES:
assessment of pain intensity | at baseline and after 8 weeks
  Participants in both groups will mark a number on a 10-cm line (0 to 10) to indicate their pain level, with 10 being the most painful. Pain ratings during exercise was assessed at baseline (pre-treatment) and after 8 weeks of treatment (post-treatment) using visual analogue numeric pain scale

SECONDARY OUTCOMES:
assessment of shoulder flexion range of motion | at baseline and after 8 weeks
  Shoulder range of motion (ROM) was assessed using a digital goniometer with participants seated. They will remove clothing from the affected shoulder and perform maximal active ROM during assessments. For shoulder flexion, the goniometer's axis will be placed over the acromion process, the stationary arm aligned with the midaxillary line, and the moving arm positioned along the central line of the upper arm.
Assessment of shoulder external rotation range of motion | at baseline and after 8 weeks
  Shoulder range of motion (ROM) was assessed using a digital goniometer with participants seated. They will remove clothing from the affected shoulder and perform maximal active ROM during assessments. External rotation is assessed when the upper limb is in a 90° abducted position. The goniometer's axis is positioned at the olecranon process, the stationary arm is aligned parallel to the ground, and the moving arm is adjusted to the ulna.
Assessment of the shoulder abduction range of motion | at baseline and after 8 weeks
  Shoulder range of motion (ROM) was assessed using a digital goniometer with participants seated. They will remove clothing from the affected shoulder and perform maximal active ROM during assessments. Shoulder abduction measurement involves positioning the goniometer's axis over the acromion process, aligning the stationary arm parallel to the spine, and setting the moving arm along the central line of the upper arm, following the protocol recommended by Lee and Kim
assessment of upper limb function | at baseline and after 8 weeks
  The study assessed upper limb function using the Arabic version of the Quick Disabilities of the Arm, Shoulder and Hand-9 scale before and after 8 weeks of treatment. The scale consists of 9 items rated on a 4-point Likert scale, where higher scores indicate increased disability and reduced function. A scaled score is computed from the total scores (0-100) using a specific formula, accommodating missing items by averaging remaining scores. Progress was measured by calculating the percent improvement in Quick Disabilities of the Arm, Shoulder and Hand-9 scores post-treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr El Ainy Learning Hospital and National Cancer Institute, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No